CLINICAL TRIAL: NCT03135860
Title: Exploratory Study to Assess the Effect of Pulsed Inhaled Nitric Oxide on Functional Respiratory Imaging Parameters in Subjects With WHO Group 3 Pulmonary Hypertension Associated With Chronic Obstructive Pulmonary Disease (COPD) on Long Term Oxygen Therapy (LTOT).
Brief Title: Effect iNO on Functional Respiratory Imaging in Subjects With WHO Group 3 Pulmonary Hypertension With COPD on Oxygen
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: This was an exploratory open-label study and has met its initial objectives
Sponsor: Bellerophon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PULSE-COPD-007
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2017-09

CONDITIONS: COPD; Pulmonary Hypertension; Chronic Obstructive Pulmonary Disease
Keywords: Inhaled Nitric Oxide; COPD; Chronic Obstructive Pulmonary Disease; Idopathic Pulmonary Fibrosis; Long Term Oxygen Therapy (LTOT)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary | interventions — Inosine

STUDY DESIGN:
Intervention Model Description: Exploratory Single Arm Study
Oversight: Data Monitoring Committee: Yes | US Export: Yes

ARMS (1):
- Inhaled Nitric Oxide 30mcg/kg/IBW/hr (Experimental): Inhaled nitric oxide 30 mcg/kg IBW/hr NO will be administered through the InoPulse Device open label for 4 weeks
  Interventions: Drug: Inhaled Nitric Oxide 30mcg/kg IBW/hr

INTERVENTIONS:
Drug: Inhaled Nitric Oxide 30mcg/kg IBW/hr — Inhaled Nitric Oxide 30 mcg/kg IBW/hr will be administered through the INOPulse Device open label for 4 weeks
  Other Names: iNO, NO,

SUMMARY:
The objective of this exploratory study is to examine the utility of high resolution computed tomography (HRCT) to measure changes in functional pulmonary imaging parameters as a function of long term iNO administrationusing the device INOpulse for 4 weeks in relation to Patient Reported Outcome (PRO) and exercise tolerance in subjects with WHO Group 3 PH associated with COPD on LTOT.

Changes from baseline to 4 weeks of pulsed iNO and after 2 weeks of withdrawal from pulsed iNO will be evaluated.

DETAILED DESCRIPTION:
In this study, pulmonary hypertension (PH) is defined as systolic pulmonary arterial pressure (sPAP) ≥ 38 mmHg by 2-D echocardiogram with Doppler.

NO cylinder concentrations (4880 ppm) at a dose of 30 mcg/kg Ideal Body Weight (IBW)/hr (INOpulse setting of 30 mcg/kg IBW/hr) will be administered.

During the screening visit all the inclusion and exclusion criteria will be checked. Eligible patients will return to the site for visit 1. During visit 1 baseline HRCT scans with contrast agent will be obtained at Functional Residual Capacity (FRC) and Total Lung Capacity (TLC). Before the scans are taken a urine pregnancy test will be obtained in female patients with childbearing potential. A retest of the eGFR CKD-EPI value should also be performed before administering the contrast agent, if there is a clinical indication according to the investigator. The treatment will be started after all baseline assessments (physical examination, patency of nares, eGFR CKD-EPI determination, urine pregnancy test, HRCT scans, vital signs including oxygen saturation measurement, Electrocardiogram (ECG), Arterial Blood Gas (ABG), MetHb, 6-minutes walking distance (6MWD) (before and after the 6 MWD a Borg Category Ratio (Borg CR10) leg fatigue and dyspnea scale will be executed and during the 6MWD the oxygen saturation will be measured), PRO, spirometry). A second TLC and FRC scan with contrast agent during the iNO treatment will be taken. The scans will be taken whilst the patient is under iNO treatment for at least 20 minutes on the iNOpulse specific cannula. After the scans taken during the iNO treatment are performed some of the baseline assessments will be repeated whilst the patient is on iNO treatment (vital signs including oxygen saturation measurement, ABG, MetHb, 6MWD (before and after the 6 MWD a Borg CR10 leg fatigue and dyspnea scale will be executed and during the 6MWD the oxygen saturation will be measured), PRO, spirometry). During visit 1 the investigator will discontinue iNO to assess if rebound pulmonary hypertension occurs. In the first 2 patients, iNO therapy will be discontinued while 2D echo is performed to assess sPAP. Furthermore, NIBP, HR, SpO2 will be measured. In the remaining patients the following additional safety assessments (NIBP, HR, SpO2) will be performed while the patient is discontinued at least 20 minutes of iNO. If the investigator considers it is safe to restart the iNO-therapy, the patient will start chronic iNO treatment. After the results of the safety assessments of the 2 first patients are collected a safety meeting will be held to evaluate the results. Depending on the results, the additional 2D echo may be performed in additional patients. Subjects will be contacted via telephone or e-mail ± 24 hours after visit 1, for assessment of vital status, concomitant medications and the occurrence of new AEs or worsening of previously existing recorded AEs and PRO (= visit 2). After 2 weeks of treatment of iNO with a dosage of 30 mcg/kg IBW/hr during at least 12 hours a day patients will be asked to return to the site for visit 3. During that visit following measurements will be performed: patency of nares will be checked, vital signs including oxygen saturation measurement, MetHb, 6MWD (with Borg CR10 leg fatigue and dyspnea scale and oxygen saturation measurement), PRO and AE assessment. After 4 weeks treatment visit 4 will be conducted. 2D - echocardiogram with Doppler (immediately after the 2D - echocardiogram with Doppler NIBP, HR, SpO2 will be measured) and HRCT scans with contrast agent under iNO pulse will be taken. Before the scans are taken an urine pregnancy test will be obtained, if applicable. A retest of the eGFR CKD-EPI value should also be performed before administering the contrast agent, if there is a clinical indication according to the investigator. Spirometry assessments will be performed, patency of nares, ECG, ABG, MetHb, 6MWD (with Borg CR10 fatigue and dyspnea scale and oxygen saturation measurement), PRO will be assessed. After all assessments are completed, iNO will be discontinued. Twenty minutes after discontinuation of iNO-therapy, spirometry, PRO, MetHb, 6MWD (before and after the 6 MWD a Borg CR10 leg fatigue and dyspnea scale will be executed and during the 6MWD the oxygen saturation will be measured) and 2D-echocardiogram with Doppler measurements measurement will be repeated. Vital signs with oxygen saturation will be measured immediately after the 2D-echocardiogram with Doppler. After all the assessments the patient is placed back on his/her prescribed dose of LTOT using their usual cannula. The patient will be assessed for any signs of acute withdrawal. Therefore vital signs including oxygen saturation will be measured.

At visit 5, two weeks after discontinuation of iNO treatment repeat vital signs with oxygen saturation measurement, physical examination, patency of nares, spirometry, 2D-echocardiogram with Doppler (immediately after the 2D - echocardiogram with Doppler NIBP, HR, SpO2 will be measured), ABG, MetHb, 6MWD(with Borg CR10 leg fatigue and dyspnea scale and oxygen saturation measurement), and PRO will be performed. If applicable a last urine pregnancy test will be executed to make sure no pregnancy occurred during the study. If there are no follow-up actions for a patient at this visit, it will be considered as a completion of study participation / end of study for that particular patient.

ELIGIBILITY:
Inclusion Criteria:

- 1. Male or female patient 2. A confirmed diagnosis of COPD by the Global initiative for chronic Obstructive Lung Disease (GOLD) criteria 3. Pulmonary hypertension will be defined as sPAP ≥ 38 mmHg as determined by echocardiogram (not obtained within ± 7 days of an exacerbation) within the past 12 months.

4. Current or former smokers with at least 10 pack-years of tobacco cigarette smoking before study entry 5. Age ≥ 40 years, ≤ 85 years 6. A post-bronchodilatory FEV1/FVC < 0.7 and a FEV1 < 60% predicted (values obtained within 6 months prior to screening can be used unless obtained within ± 7 days of an exacerbation; otherwise, the test must be performed during screening) 7. Receiving LTOT for ≥ 3 months and ≥ 10 hours per day as determined by history 8. Females of childbearing potential must have a negative pre-scan urine pregnancy test 9. Signed informed consent prior to the initiation of any study mandated procedures or Assessments

Exclusion Criteria:

* 1. Males who have the intention to father a child during the study. 2. A diagnosis of asthma or other non-COPD respiratory disease, in the opinion of the Investigator 3. Lack of patency of nares upon physical examination 4. Experienced during the last month an exacerbation requiring:

  1. start of or increase in systemic oral corticosteroid therapy and/or
  2. hospitalization 5. Left ventricular dysfunction as measured by:

  <!-- -->

  1. Screening echocardiographic evidence of left ventricular systolic dysfunction (left ventricular ejection fraction [LVEF] < 40%), or
  2. Screening echocardiographic evidence of left ventricular diastolic dysfunction >moderate (i.e., > Grade 3), or
  3. Any history of pulmonary capillary wedge pressure (PCWP), left atrial pressure (LAP) or left ventricular end diastolic pressure (LVEDP) > 18 mmHg as measured during cardiac catheterization within the past 6 months unless documented to have resolved by a subsequent cardiac catheterization 6. Renal impairment (i.e., an estimated GFR CKD-EPI < 30 ml/min/1.73 m2) or history of renal failure using the equation:

     Men:

     crs< 0.9 mg/dL: eGFRCKD-EPI = 141 × (crs /0.9)-0.411 × 0.993Age crs≥ 0.9 mg/dL: eGFRCKD-EPI = 141 × (crs /0.9)-1.209 × 0.993Age

     Woman:

     crs< 0.7 mg/dL: eGFRCKD-EPI = 144 × (crs /0.7)-0.329 × 0.993Age crs≥ 0.7 mg/dL: eGFRCKD-EPI = 144 × (crs /0.7)-1.209 × 0.993Age where crs= Normal and elevated serum creatinine Subjects with possible compromised kidney function (i.e., Glomerular Filtration Rate estimated using the Modification of Diet in Renal Disease equation [eGFR CKD-EPI] between 30 and 60 ml/min/1.73 m2) may be enrolled provided the Radiology Department and Principal Investigator review the medical records of subjects with an eGFR CKD-EPI between 30 and 60 ml/min/1.73 m2 in order to confirm the contrast agent can be safely administered to these subjects and approval by both the Radiology Department and Principal Investigator must be obtained before enrolling these subjects.

     7. Known allergy to contrast media. 8. Clinically significant valvular heart disease that may contribute to PH, including mild or greater aortic valvular disease (aortic stenosis or regurgitation) and/or moderate or greater mitral valve disease (mitral stenosis or regurgitation), or status post mitral valve replacement 9. Use within 30 days of screening or current use of approved PH medications such as sildenafil or bosentan (use of Cialis® or Viagra® for erectile dysfunction is permitted) 10. Use of investigational drugs or devices within 30 days prior to enrollment into the study 11. Any underlying medical or psychiatric condition that, in the opinion of the Investigator, makes the subject an unsuitable candidate for the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

PRIMARY OUTCOMES:
change in lobar blood volume at total lung capacity with iNO and the change in lobar blood volume with iNO after 4 weeks of treatment with iNO as measured by HRCT. | After 4 weeks of treatment
  The primary endpoint in this exploratory study is the change in lobar blood volume at total lung capacity with iNO and the change in lobar blood volume with iNO after 4 weeks of treatment with iNO as measured by HRCT.

SECONDARY OUTCOMES:
Blood vessel % and density on lobar level | after 4 weeks of treatment
  are the changes from baseline measured by HRCT with pulsed iNO and after dosing with pulsed iNO in Blood vessel % and density on lobar level
• Blood vessel % and density on lobal level compared among patients with emphysema, chronic bronchitis or combined emphysema and chronic bronchitis as assessed by HRCT | after 4 week of treatment
  are the changes from baseline measured by HRCT with pulsed iNO and after dosing with pulsed iNO in Blood vessel % and density on lobal level compared among patients with emphysema, chronic bronchitis or combined emphysema and chronic bronchitis as assessed by HRCT
Total lung volume at TLC | after 4 week of treatment
  the changes from baseline measured by HRCT with pulsed iNO and after dosing with pulsed iNO in Total lung Volume at TLC
Lobar volumes at TLC | after 4 weeks of treatment
  the changes from baseline measured by HRCT with pulsed iNO and after dosing with pulsed iNO in Lobar volumes at TLC
Internal airflow distribution based on lobar expansion | after 4 weeks of treatment
  the changes from baseline measured by HRCT with pulsed iNO and after dosing with pulsed iNO in Internal airflow distribution based on lobar expansion
Airway volume down to generation 8-10 at TLC | After 4 weeks of treatment
  the change in lobar blood volume at total lung capacity with iNO and the change in lobar blood volume with iNO in Airway volume down to generation 8-10 at TLC
Computational Fluid Dynamics (CFD)-based resistance on lobar level | after 4 weeks of treatment
  change in lobar blood volume at total lung capacity with iNO and the change in lobar blood volume with iNO in Computational Fluid Dynamics (CFD)-based resistance on lobar level
Ventilation/perfusion (V/Q) matching | after 4 weeks of treatment
  the change in lobar blood volume at total lung capacity with iNO and the change in lobar blood volume with iNO in Ventilation/perfusion (V/Q) matching
Spirometry | after 4 weeks of treatment
  the changes from baseline measured by HRCT with pulsed iNO and after dosing with pulsed iNO in Spirometry
Change from baseline 6MWD; Borg CR10 Dyspnea and Leg Fatigue Score ; PRO | after 4 weeks of treatment two weeks of withdrawal
  Change in baseline to 4 weeks of pulsed iNO and after 2 weeks of withdrawal from pulsed iNO in:6MWD; Borg CR10 Dyspnea and Leg Fatigue Score ; PRO
Change from baseline to 4 weeks of treatment and two weeks of withdrawal | after 4 weeks of treatment two weeks of withdrawal
  • Right Ventricular (RV) and Left Ventricular (LV) size and function, PAP as measured by 2D-echocardiogram with Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No